CLINICAL TRIAL: NCT02891070
Title: A Randomised Controlled Study to Evaluate the Efficacy and Safety of Fibrin Sealant, Vapour Heated, Solvent/Detergent Treated FS VH S/D 500 S-apr (Tisseel) Compared to DuraSeal Dural Sealant as an Adjunct to Sutured Dural Repair in Cranial Surgery.
Brief Title: Efficacy and Safety of FS VH S/D 500 S-apr (Tisseel) as an Adjunct to Sutured Dural Repair in Cranial Surgery
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Baxter Healthcare Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 3599-001; 2015-005535-40 (EudraCT Number)
Record Dates: First submitted 2016-09-01; First posted 2016-09-07 (Estimated); Results first posted 2019-09-10 (Actual); Last update posted 2019-09-10 (Actual); Status verified 2019-08

CONDITIONS: Cerebrospinal Fluid Leak
Keywords: Cranial Surgery; Cerebrospinal Fluid Leak; Tisseel
MeSH Terms: conditions — Cerebrospinal Fluid Leak | interventions — Low Density Lipoprotein Receptor-Related Protein-1; Fibrin Tissue Adhesive

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- FS VH S/D 500 s-apr (Experimental): FS VH S/D 500 s-apr (Tisseel), single use treatment, intraoperative
  Interventions: Drug: FS VH S/D 500 s-apr
- DuraSeal Dural Sealant (Active Comparator): DuraSeal Dural Sealant, single use treatment, intraoperative
  Interventions: Device: DuraSeal Dural Sealant

INTERVENTIONS:
Drug: FS VH S/D 500 s-apr
  Other Names: Tisseel
  Arms: FS VH S/D 500 s-apr
Device: DuraSeal Dural Sealant
  Arms: DuraSeal Dural Sealant

SUMMARY:
The objective of this study is to evaluate the safety and efficacy of FS VH S/D 500 s-apr for use as an adjunct to sutured dural repair in cranial surgery.

ELIGIBILITY:
Inclusion Criteria:

1. Patients undergoing craniotomy/craniectomy for pathological processes in the PF or ST region
2. Patients must be willing and able to participate in the study and provide written IC before any protocol specific assessment is performed
3. Patients must be willing to receive peri-operative antibiotic prophylaxis
4. Female patients of childbearing potential must present with a negative serum pregnancy test, and must agree to employ adequate birth control measures [restricted to abstinence, barrier contraceptives, intrauterine contraceptive devices or licensed hormonal products] for the duration of their participation in the study
5. Patients are willing and able to comply with the requirements of the protocol

Exclusion Criteria:

1. Patients with a dural lesion from a recent surgery that still has the potential for CSF leakage
2. Patients who had undergone chemotherapy treatment, excluding hormonal therapy, within 3 weeks prior to the planned procedure, or with chemotherapy scheduled within 7 days following surgery
3. Patients with radiation therapy to the surgical site or standard fractionated radiation therapy scheduled within 7 days following surgery
4. Patients with a previous craniotomy/craniectomy within 6 months prior to the study surgery
5. Use of corticosteroids on a chronic basis (defined as daily use of corticosteroids for ≥8 weeks) for purposes other than decreasing the symptoms of systemic chemotherapy (unless if those steroids were discontinued 4 weeks prior to the planned surgery)
6. Patients with a known hypersensitivity to the components of the IP or control (human fibrinogen, synthetic aprotinin, human albumin, human FXIII, tri sodium citrate, histidine, niacinamide, polysorbate 80, human thrombin, polyethylene glycol [PEG], trilysine amine)
7. Patients with a known hypersensitivity to US Federal Drug & Cosmetic Blue #1 dye
8. Evidence of an infection indicated by any one of the following: clinical examination supporting the diagnosis of infection, fever (temperature >100.7°F or 38.2°C), positive urine culture, positive blood culture, positive chest X ray consistent with pulmonary infection, or infection along the planned surgical path. A white blood cell (WBC) count of <20000 cells/µL is permitted if the patient is being treated with steroids in the absence of all other infection parameters
9. Female patients of childbearing potential with a positive pregnancy test or intent to become pregnant during the clinical study period
10. Female patients who are nursing
11. Patients with exposure to another investigational drug or device clinical trial within 30 days prior to enrolment or anticipated in the 60-day Follow-up period
12. Patients with severely altered renal function as confirmed by local laboratory reference ranges for serum creatinine and/or hepatic function (alanine aminotransferase [ALT], aspartate aminotransferase >3 × upper limit of normal [ULN])
13. Patients who currently have or have had a compromised immune system (such as Acquired Immune Deficiency Syndrome [AIDS]) or autoimmune disease, or were on chronic immunosuppressant agents
14. Patients with uncontrolled diabetes as evidenced by the institution's standard of care (glycated haemoglobin [HbA1c] >7%, blood glucose, etc.)
15. Patients with traumatic injuries to the head
16. Patients with dural injury during craniotomy/craniectomy that cannot be eliminated by widening the craniotomy/craniectomy to recreate the native dural cuff
17. Patients requiring surgical approaches that would not allow sutured dural closure such as trans-sphenoidal or translabyrinthine/-petrosal/-mastoid. Superficial penetration of mastoid air cells is allowed
18. Patients with hydrocephalus, except occlusive hydrocephalus caused by PF pathology or incompletely open cerebrospinal fluid pathways, to be treated during surgical procedure
19. Existing CSF (ventricular, etc.) drains, Cushing/Dandy cannulation, or Burr holes which damage the dura
20. Patients with confined bony structures where nerves are present and neural compression may result due to swelling

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 224 (Actual)
Dates: Start 2016-10-11 (Actual); Primary Completion 2018-08-22 (Actual); Study Completion 2018-08-22 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Qing Li, MD, PhD, Study Director — Baxter Healthcare
Locations (25):
- United States (10):
  - Southern Illinois University School of Medicine, Springfield, Illinois
  - Baystate Medical Center, Springfield, Massachusetts
  - Henry Ford Hospital, Detroit, Michigan
  - University of Minnesota, Minneapolis, Minnesota
  - University Hospitals Case Medical Center, Cleveland, Ohio
  - The Ohio State University, Columbus, Ohio
  - Temple University School of Medicine, Philadelphia, Pennsylvania
  - University of Pittsburgh Medical Center, Pittsburgh, Pennsylvania
  - Houston Methodist Neurological Institute, Houston, Texas
  - University of Virginia School of Medicine, Charlottesville, Virginia
- Czechia (6):
  - University Hospital Brno, Brno
  - St. Anne's University Hospital Brno, Brno
  - University Hospital Hradec Kralove, Hradec Králové
  - University Hospital Ostrava, Ostrava
  - Hospital Na Homolce, Prague
  - University Hospital Motol, Praha 5 - Motol
- Germany (3):
  - University Hospital Leipzig, Leipzig
  - Hospital Bogenhausen Municipal Hospital, Munich
  - University Hospital Rostock, Rostock
- Spain (6):
  - University Hospital Germans Trias I Pujol, Badalona
  - Hospital Clinic I Provincial de Barcelona, Barcelona
  - University Hospital Foundation Jimenez Diaz, Madrid
  - University Hospital 12 de Octubre, Madrid
  - University Hospital Son Espases, Palma de Mallorca
  - University General Hospital of Valencia, Valencia

RESULTS

PARTICIPANT FLOW:
Groups:
- Tisseel: Tisseel (FS VH S/D 500 s-apr), single use treatment, was administered intra-operatively with sutures during dural closure. Product was applied with cannula by dripping in a thin and continuous layer with a 5 mm overlap on each side of the sutured line, ensuring that all suture holes were covered.
- DuraSeal: DuraSeal Dural Sealant, single use treatment, was administered intra-operatively with sutures during dural closure. The product was applied with the DuraSeal System Applicator by spraying a thin (1 - 2 mm) coating, ensuring that all suture holes were covered.
Period: Overall Study
Arm/Group | Tisseel | DuraSeal
Started | 110 | 114
Completed | 100 | 106
Not Completed | 10 | 8
Not completed — Adverse Event | 1 | 0
Not completed — Physician Decision | 0 | 1
Not completed — Lost to Follow-up | 4 | 4
Not completed — Other | 1 | 0
Not completed — Protocol Violation | 0 | 1
Not completed — Withdrawal by Subject | 1 | 2
Not completed — Death | 3 | 0

BASELINE CHARACTERISTICS:
Population: Full analysis set (FAS): The FAS consisted of all patients who were randomized and treated with at least 1 dose of IP/control. Patients were analyzed as randomized.
Groups:
- Total: Total of all reporting groups
Arm/Group | Tisseel | DuraSeal | Total
Number analyzed (Participants) | 110 | 114 | 224
Age, Continuous [Mean (Standard Deviation); unit: Years] | 51.8 (14.24) | 51.3 (14.85) | 51.5 (14.53)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 66 | 65 | 131
  Male | 44 | 49 | 93
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 2 | 2 | 4
  White | 97 | 101 | 198
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 11 | 11 | 22

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With No CSF Leak During and After Surgery
Description: Participants who have no intra-operative CSF leak from dural repair after up to two applications during Valsalva maneuver (25 cm H2O for up to 5 - 10 seconds), or post-operative CSF leak within 30 (+3) days post-operatively. The Valsalva maneuver was performed by the anaesthesiologist to increase the intra-thoracic pressure (e.g., by increasing the positive end-expiratory pressure or by giving a large tidal volume and holding the inflating pressure) to approximately 25 cm H2O, constantly for up to 5 - 10 seconds to transiently elevate the intracranial pressure and test for any CSF leaks. The suture line was to be watertight after up to two product/control applications and Valsalva maneuvers.
Time Frame: Day 0 (Intra-operative) to Day 30 (+/-3 days) post-operative
Population: Per-protocol analysis set (PPS): The PPS was defined as a subset of the FAS. Patients with any major deviation that may have impacted the primary efficacy parameter were excluded from the PPS.
Measure: Count of Participants; unit: Participants
Arm/Group | Tisseel | DuraSeal
Number analyzed (Participants) | 89 | 95
Participants | 76 | 87
Statistical Analysis 1: Comparison: Tisseel vs DuraSeal; Test type: Non-Inferiority — To demonstrate non-inferiority (NI) of Tisseel to DuraSeal for the primary endpoint, the lower limit of the 95% CI (based on normal approximation) for the difference in average predicted proportions had to be greater than -10%; Regression, Logistic; Mean Difference (Net) = -9.29, 95% CI 2-sided [-21.11 to 2.54] — Difference in Average Predicted Proportion (Tisseel - Duraseal)

2. Secondary Outcome: Number of Participants With no Intra-operative CSF Leaks Following Final Valsalva Maneuver
Description: Assessment of whether the suture line was not watertight causing CSF leaks after up to two product/control applications and Valsalva maneuvers.
Time Frame: Day 0 (Intra-operative)
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Tisseel | DuraSeal
Number analyzed (Participants) | 89 | 95
Participants | 89 | 95

3. Secondary Outcome: Number of Participants With CSF Leaks Within 30 (+3) Days Post-operatively
Description: Cerebrospinal fluid leak was defined as any overt flow, seepage, weeping, or sweating of CSF through the dura suture line, regardless of volume. All post-operative CSF leaks were primarily diagnosed based on a detailed history and physical examination, including neurological examination. Although not standard of care post-operatively, imaging tests such as computed tomography/magnetic resonance imaging (MRI) were considered if there was a high clinical suspicion of a CSF leak.
Time Frame: Day 0 (Intra-operative) to Day 30 (+/-3 days) post-operative
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Tisseel | DuraSeal
Number analyzed (Participants) | 89 | 95
Participants | 8 | 2
Statistical Analysis 1: Comparison: Tisseel vs DuraSeal; Test type: Other; Regression, Logistic; Mean Difference (Net) = -9.29, 95% CI 2-sided [-21.11 to 2.54] — Difference in Average Predicted Proportion (Tisseel - Duraseal)

4. Secondary Outcome: Duration in Surgery (Minutes)
Description: Patients undergoing elective cranial surgery for the treatment of a pathological condition (e.g., benign/malignant tumours, vascular malformations, or Chiari type 1 malformations) specifically located in the posterior fossa (PF) or supratentorial (ST) regions.
Time Frame: Day 0 (intra-operatively)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Minutes
Arm/Group | Tisseel | DuraSeal
Number analyzed (Participants) | 89 | 95
Minutes | 241.8 (100.80) | 210.3 (90.49)
Statistical Analysis 1: Comparison: Tisseel vs DuraSeal; Test type: Other; p = 0.0241, Wilcoxon (Mann-Whitney)

5. Secondary Outcome: Time From Dural Closure (Application of IP) Until End of Surgery
Description: Suture closure techniques include continuous simple, continuous locked, interrupted.
Time Frame: Day 0 (Intra-operatively)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Minutes
Arm/Group | Tisseel | DuraSeal
Number analyzed (Participants) | 89 | 95
Minutes | 34 (16.13) | 31.4 (17.07)
Statistical Analysis 1: Comparison: Tisseel vs DuraSeal; Test type: Other; p = 0.1015, Wilcoxon (Mann-Whitney)

6. Secondary Outcome: Length of Stay in Hospital (Days).
Description: Days in hospital calculation is Day 0 - Discharge.
Time Frame: Day 0 to Day 60 (Study Completion)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | Tisseel | DuraSeal
Number analyzed (Participants) | 89 | 95
Days | 13.5 (15.57) | 12.6 (8.67)
Statistical Analysis 1: Comparison: Tisseel vs DuraSeal; Test type: Other; p = 0.9943, Wilcoxon (Mann-Whitney)

7. Post Hoc Outcome: Number of Surgical Site Infections (SSI)
Description: Surgical site infections were evaluated by the surgeon or designated physician according to United States (US) National Healthcare Safety Network (NHSN) criteria as specified in the study protocol.
Time Frame: Day 0 (Intra-operative) to Day 30 (+/-3 days) post-operative
Population: Safety analysis set (SAS): The SAS consisted of all patients who were treated with IP/Control. Patients were analyzed as treated.
Measure: Number; unit: SSI
Arm/Group | Tisseel | DuraSeal
Number analyzed (Participants) | 110 | 114
SSI | 1 | 4
Statistical Analysis 1: Comparison: Tisseel vs DuraSeal; Test type: Other; Regression, Logistic; Mean Difference (Net) = -5.11, 95% CI 2-sided [-13.60 to 3.39]

ADVERSE EVENTS:
Time Frame: Day -30 (Pre-operative) to Day 60 (+/- 3 days)
Description: Treatment-Emergent Adverse Events (TEAE) were reported for both Adverse Event (AE) and Serious Adverse Events (SAE). TEAE's are events that began or worsen in severity after the first administration of treatment.
Arm/Group | Tisseel | DuraSeal
All-Cause Mortality (participants affected / at risk) | 3/110 | 0/114
Serious Adverse Events (participants affected / at risk) | 22/110 | 17/114
Other Adverse Events (participants affected / at risk) | 46/110 | 46/114
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Tisseel (N=110) | DuraSeal (N=114)
Cardiac Arrest (Cardiac disorders) | 1 (1) | 0 (0)
Adrenal Insufficiency (Endocrine disorders) | 1 (1) | 0 (0)
Abdominal Discomfort (Gastrointestinal disorders) | 0 (0) | 1 (1)
Pyrexia (General disorders) | 1 (1) | 0 (0)
Brain Abscess (Infections and infestations) | 0 (0) | 2 (2)
Brain Empyema (Infections and infestations) | 0 (0) | 1 (1)
Epidural Empyema (Infections and infestations) | 0 (0) | 1 (1)
Hepatitis E (Infections and infestations) | 1 (1) | 0 (0)
Osteomyelitis (Infections and infestations) | 0 (0) | 2 (2)
Pneumonia (Infections and infestations) | 1 (1) | 1 (1)
Soft Tissue Infection (Infections and infestations) | 0 (0) | 1 (1)
Wound Infection (Infections and infestations) | 0 (0) | 2 (2)
Brain Contusion (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Extradural Haematoma (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Femur Fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Pneumocephalus (Injury, poisoning and procedural complications) | 1 (2) | 0 (0)
Post Procedural Haemorrhage (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Pseudomeningocele (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Wound Dehiscence (Injury, poisoning and procedural complications) | 0 (0) | 2 (2)
Wound Haematoma (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Brain Oedema (Nervous system disorders) | 1 (1) | 2 (2)
Cerebrospinal Fluid Leakage (Nervous system disorders) | 7 (7) | 1 (1)
Dizziness (Nervous system disorders) | 1 (1) | 0 (0)
Hydrocephalus (Nervous system disorders) | 3 (3) | 1 (1)
Idiopathic Intracranial Hypertension (Nervous system disorders) | 0 (0) | 1 (1)
Sensorimotor Disorder (Nervous system disorders) | 0 (0) | 1 (1)
Superior Sagittal Sinus Thrombosis (Nervous system disorders) | 0 (0) | 1 (1)
Thalamic Infarction (Nervous system disorders) | 1 (1) | 0 (0)
Aspiration (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Pulmonary Embolism (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Respiratory Distress (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Tisseel (N=110) | DuraSeal (N=114)
Constipation (Gastrointestinal disorders) | 8 (9) | 5 (5)
Nausea (Gastrointestinal disorders) | 10 (12) | 14 (16)
Vomiting (Gastrointestinal disorders) | 10 (15) | 14 (17)
Pain (General disorders) | 15 (15) | 15 (16)
Pyrexia (General disorders) | 3 (6) | 7 (7)
Dizziness (Nervous system disorders) | 6 (8) | 3 (4)
Headache (Nervous system disorders) | 20 (25) | 21 (25)
Hypertension (Vascular disorders) | 5 (5) | 6 (6)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2017-11-06): https://cdn.clinicaltrials.gov/large-docs/70/NCT02891070/Prot_000.pdf
  • Statistical Analysis Plan (2017-08-10): https://cdn.clinicaltrials.gov/large-docs/70/NCT02891070/SAP_001.pdf